CLINICAL TRIAL: NCT01583335
Title: Prevention of Weight Gain Among Normal Weight, Obesity Susceptible, Pre-school Children - a Randomized Controlled Interventions Study.
Brief Title: The Healthy Start Project: Primary Prevention of Overweight in Preschool Children Susceptible to Future Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); The Danish Medical Research Council (Other); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Berit Lilienthal Heitmann, Professor, Ph.D., Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Tryg-7984-07
Record Dates: First submitted 2012-03-31; First posted 2012-04-24 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Susceptibility; Prevention; Diet; Physical activity; Sleep; Family stress
MeSH Terms: conditions — Overweight; Obesity; Disease Susceptibility; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Improved lifestyle (Experimental)
  Interventions: Behavioral: Lifestyle habits, including sleep and stress
- Control group (No Intervention): The control group was seen at baseline and follow-up, but not in between.
- Shadow group (No Intervention): The shadow group was followed in registers exclusively

INTERVENTIONS:
Behavioral: Lifestyle habits, including sleep and stress — The intervention group was offered up to 10 individual consultations focusing on improving diet, physical activity and sleep habits and reducing stress. Moreover, the intervention group was offered participation in monthly cooking classes and playing arrangements
  Arms: Improved lifestyle

SUMMARY:
Obesity prevention should remain a priority, although there is some evidence of a possible leveling off in some age groups across European countries and in USA, Japan and Australia. Besides adult health problems such as type-2 diabetes and cardiovascular diseases, obesity in childhood is associated with psychological and social problems, low self-esteem, stigmatization and being teased and bullied by friends. Danish research suggests that the causes behind the increase in obesity occurrence are present already in early childhood, and that prevention of obesity therefore has to start early. Research has suggested that at least three sub-groups can be considered susceptible to develop obesity: Children with obesity among their 1st degree relatives; children with a high birth weight or children coming from socially disadvantaged families (low socioeconomic status). Earlier intervention programs has showed little effect in preventing excessive weight gain and knowledge on how to develop effective intervention programs that reduce overweight and obesity remains limited. It has been suggested that future prevention programs may be more successful if specifically targeting groups that are at high risk, as mention above, of excessive weight gain.

Based on these suggestions, the "Sund Start" project was initiated. The purpose of the study was to determine whether aiming prevention towards 2-6 years old Danish children who were yet normal weight, but were considered susceptible to develop overweight or obese could prevent later on risk of becoming overweight or obese. Furthermore, to investigate if it was possible to improve diet habits, increase physical activity, reduce stress and improve sleeping habits among children at high risk for later on overweight and obesity.

The "Sund Start" project will contribute with knowledge about whether targeting normal weight, predisposed children is effective in preventing overweight and obesity, and if reduced stress and improved sleep, should be considered important new obesity prevention tools. Moreover, the project will contribute with knowledge about how to change lifestyle and its effects on development of overweight and obesity in high risk Danish preschool children.

DETAILED DESCRIPTION:
In 2009, data on all births between 2004 and 2007 in 11 selected municipalities from the greater Copenhagen area was obtained from the Danish national birth register at the National Board of Health. This register contains information on all births, whether at hospital or home, on factors such as birth weight and length, height and pre-pregnant weight of the mother, parity, and Central Personal Registry number (CPR-number). Data on socioeconomic status was obtained from the administrative birth forms. This was done manually using the CPR-numbers obtained from the birth register.

After selection of the children eligible for participation, the children were allocated to three groups, (intervention group, control group, shadow group) using computer based randomization. All siblings were allocated to the same group. After the random allocation, children from the intervention group and the control group were sent a letter with an invitation to participate in the project. Children from the shadow group were also identified, and their general practitioners were contacted and asked for information on each child's height and weight.

ELIGIBILITY:
Inclusion Criteria:

* Born between 2004-2007
* Born in 11 selected municipalities in the greater Copenhagen area
* Classified as susceptible to overweight and obesity (At least one of the following risk factors present: A high birth weight (> 4000 grams), maternal pre-pregnancy obesity (BMI > 28 kg/m^2), or maternal low education (<= 10 years)
* Normal weight at baseline examination

Exclusion Criteria:

* Moved to another municipality after birth,
* Had requested protection from participation in statistical or scientific surveys based on data delivered from the Danish Central Person Registry
* No permanent address
* Lived in a children's home
* Had died
* Had emigrated
* Registered in the Danish Central Person Registry as being disappeared or had unknown life status
* Not speaking Danish
* Overweight (including obesity) at baseline examination

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1202 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | 1.3 years
  Changes between baseline and 1.3 years follow.up per intervention year in:
  Height in cm Weight in kg BMI in kg/m^2 BMI z-score in SD Waist circumference in cm Hip circumference in cm Sum of four skinfolds (biceps, triceps, subscapular and suprailiac) in cm Body composition measured by bio-electrical impedance
Anthropometric measurements | 5 years
  Changes between baseline and 5 years follow.up per intervention year in:
  Height in cm Weight in kg BMI in kg/m^2 BMI z-score in SD
Anthropometric measurements | 10 years
  Changes between baseline and 10 years follow.up per intervention year in:
  Height in cm Weight in kg BMI in kg/m^2 BMI z-score in SD

SECONDARY OUTCOMES:
Dietary intake | 1.3 years
  Four day dietary record completed Wednesday-Saturday
Priority of serving fruit and vegetables | 1.3 years
  How high do you prioritize that fruit and vegetables are served at the meals? (Scale from 1 to 4, 1 being low and 4 being high. Higher values considered better outcome)
Physical activity | 1.3 years
  Children's Physical Activity Questionnaire (C-PAQ. 7-day recording of sports, games and leisure time activities outside daycare. The response options were indicated by doing a particular activity ("yes" or "no") and by an indication of total time used on the activity during the week (minutes per week). All minutes per week were summed to obtain an indication of overall physical activity level. Higher values considered better outcome)
Sleep duration | 1.3 years
  7 day sleep record from completed questionnaire (average number of minutes sleep summed from 7 day record on sleep- and wake time points)
Child stress level | 1.3 years
  Measured concentration of cortisol in hair samples
Parental stress level | 1.3 year
  Measured concentration of cortisol in hair samples
Sleep quality | 1.3 year
  Child's sleep is considered (calm all night, a little disturbed, disturbed with occasional awakenings, very disturbed with several awakenings. Calm all night considered best outcome).
Child stress level | 1.3 year
  Strengths and Difficulties Questionnaire (SDQ). Scored 0-2 and summed to Total Difficulties score (0-40, lower score indicate better outcome), and Prosocial Behavior score (0-10, lower score indicate worst outcome)
Parental stress level | 1.3 years
  Modified version of the Swedish Parental Stress Index (PSI). Each question was scored between 0 and 2 (0 considered best score and 2 the worst), according to its estimated indication of an overall stress level. Analysis of intercorrelations among the 10 questions and a principal component analysis suggested that 9 of the 10 questions could be added together to get a score for the overall family stress level (0-18)
Daily physical activity: Enjoys being active | 1.3 years
  If the child enjoyed being physically active (Never, often, some times, usually, always. Always considered best outcome)
Meal habits: Eating breakfast together | 1.3 years
  How many times per week does the family eat breakfast together (None, 1 day, 2-3 days, 4-5 days, 6-7 days. 6-7 days considered best outcome).
Meal habits: Eating dinner together | 1.3 years
  How many times per week does the family eat dinner together (None, 1 day, 2-3 days, 4-5 days, 6-7 days. 6-7 days considered best outcome).
Meal habits: Mealtime situation | 1.3 years
  How would you describe the meals with the child (Very conflictive, little conflictive, very cozy, little cozy, don't know. Very cozy considered best outcome).
Meal habits: Pickiness | 1.3 years
  How would you describe your child's way of eating (Picky, open to new tastes, eats everything. Eats everything considered best outcome).
Meal habits: Appetite | 1.3 years
  How would you describe your child's appetite (Too big appetite, good appetite, normal appetite, too small appetite, don't know. Normal appetite considered best outcome).
Sleep quality: Difficulties falling asleep | 1.3 years
  Difficulties falling asleep (yes/no. No considered best outcome)
Sleep quality: Difficulties waking up | 1.3 years
  Difficulties waking up (yes/no. No considered best outcome)
Sleep quality: Sleep onset latency | 1.3 years
  Sleep onset latency (numerical. Lower values considered better outcome)
Sleep quality: Bedtime routines | 1.3 years
  Routine activities before bedtime (No, < 1/week, 1-2 times/week, 3-4 times/week, 5-6 times/week, every day. Every day considered best outcome)
Sleep quality: Joining parents' bed | 1.3 years
  Child joining parents' bed (yes/no. If yes, how often (< 1/month, 1-3 times/month,1-3 times/week, 4-6 times/week, every night)
Sleep quality: Falling asleep | 1.3 years
  Child afraid to fall asleep (Never, rarely, some times, often, very often. Never considered best outcome)
Sleep quality: Dreams | 1.3 years
  Child has frightening/upsetting dreams (Never, rarely, some times, often, very often. Never considered best outcome)
Daily physical activity: Means of transportation | 1.3 years
  Means of transportation to and from day-care, and frequency (Walk, strolling, bike on its own, biked by parent, and bus, train or car, number of times per week (1,2,3,4 or 5. Walking or biking on its own considered best outcome).
Daily physical activity: Activity compared to other children | 1.3 years
  How active is the child compared to other children at similar age? (as active, somewhat active, very active, don't know. Very active considered best outcome)
Daily physical activity: Activity with parents | 1.3 years
  Frequency of which one or both parents were physically active with the child (once per week, 2-4 times per week, 5-7 times per week, multiple times per day. Multiple times per day considered best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Berit L Heitmann, Professor, Study Director — Parker Institute
Locations (1):
- Parker Institute, Research Unit for Dietary Studies, Frederiksberg, Denmark

REFERENCES:
- [Derived] Rohde JF, Larsen SC, Handel MN, Olsen NJ, Stougaard M, Heitmann BL. Associations between Parental Stress and Subsequent Changes in Dietary Intake and Quality among Preschool Children Susceptible to Obesity. Int J Environ Res Public Health. 2021 Mar 30;18(7):3590. doi: 10.3390/ijerph18073590. PMID 33808371
- [Derived] Zheng M, Rangan A, Olsen NJ, Heitmann BL. Longitudinal association of nighttime sleep duration with emotional and behavioral problems in early childhood: results from the Danish Healthy Start Study. Sleep. 2021 Jan 21;44(1):zsaa138. doi: 10.1093/sleep/zsaa138. PMID 32691048
- [Derived] Olsen NJ, Rohde JF, Handel MN, Stougaard M, Mortensen EL, Heitmann BL. Joining Parents' Bed at Night and Overweight among 2- to 6-Year-Old Children - Results from the 'Healthy Start' Randomized Intervention. Obes Facts. 2018;11(5):372-380. doi: 10.1159/000492003. Epub 2018 Oct 12. PMID 30308484
- [Derived] Handel MN, Larsen SC, Rohde JF, Stougaard M, Olsen NJ, Heitmann BL. Effects of the Healthy Start randomized intervention trial on physical activity among normal weight preschool children predisposed to overweight and obesity. PLoS One. 2017 Oct 9;12(10):e0185266. doi: 10.1371/journal.pone.0185266. eCollection 2017. PMID 28991907
- [Derived] Olsen NJ, Buch-Andersen T, Handel MN, Ostergaard LM, Pedersen J, Seeger C, Stougaard M, Traerup M, Livemore K, Mortensen EL, Holst C, Heitmann BL. The Healthy Start project: a randomized, controlled intervention to prevent overweight among normal weight, preschool children at high risk of future overweight. BMC Public Health. 2012 Aug 1;12:590. doi: 10.1186/1471-2458-12-590. PMID 22852799
- See also: Click here for latest information about the "Sund Start" study. — http://www.sundstart.nu